CLINICAL TRIAL: NCT06768775
Title: The Impact of Pastured Livestock Food Consumption on Fatty Acid and Metabolomic Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephanvanvliet, Assistant Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14156
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Omega 3 Fatty Acids
Keywords: Regenerative agriculture; Conventional farming; Fatty acid profiles; Omega-3; Inflammatory markers; Metabolomics; Pastured meat; Nutritional biomarkers; Diet intervention; Human health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pastured Livestock Products Group (Experimental): Participants in this group will consume meat and eggs sourced from regenerative/pastured farming practices. Weekly allocations include chicken (300-500g), beef (500-700g), pork (300-500g), and 8-12 eggs, depending on the habitual caloric intake of participants. These products are provided for the 16-week intervention, with adherence monitored through dietary logs and 24-hour recalls.
  Interventions: Dietary Supplement: Pastured Livestock Diet
- Conventional Livestock Products Group (Experimental): Participants in this group will consume meat and eggs sourced from conventional farming practices. Weekly allocations include chicken (300-500g), beef (500-700g), pork (300-500g), and 8-12 eggs, depending on the habitual caloric intake of participants. These products are provided for the 16-week intervention, with adherence monitored through dietary logs and 24-hour recalls.
  Interventions: Dietary Supplement: Conventional Livestock Diet

INTERVENTIONS:
Dietary Supplement: Pastured Livestock Diet — Participants will consume a diet consisting of animal-source foods (chicken, beef, pork, and eggs) from regenerative/pastured farming practices. Foods will be provided weekly in specific quantities for a 16-week intervention. Adherence will be monitored through dietary logs and ASA24 dietary assessments.
  Arms: Pastured Livestock Products Group
Dietary Supplement: Conventional Livestock Diet — Participants will consume a diet consisting of animal-source foods (chicken, ground, pork, and eggs) from conventional farming practices. Foods will be provided weekly in specific quantities for a 16-week intervention. Adherence will be monitored through dietary logs and ASA24 dietary assessments.
  Arms: Conventional Livestock Products Group

SUMMARY:
The goal of this clinical trial is to evaluate the effects of consuming meat and eggs from regenerative/pastured versus conventional farming practices on health biomarkers in middle-aged adults. The main questions it aims to answer are:

How does consumption of pastured animal products influence red blood cell omega-3 fatty acid levels, inflammatory markers, and metabolomic profiles compared to conventional animal products?

What are the potential metabolic health benefits or risks associated with consuming animal products from regenerative farming practices?

Researchers will compare participants consuming pastured meat and eggs to those consuming conventional meat and eggs to determine differences in health outcomes.

Participants will:

Consume study-provided chicken thighs, ground beef, ground pork, and eggs for 16 weeks.

Attend clinic visits for blood, urine, and stool sample collection before and after the intervention.

Complete dietary assessments to monitor compliance.

DETAILED DESCRIPTION:
This randomized, double-blind, parallel-arm clinical trial investigates the impact of consuming animal products from regenerative/pastured versus conventional farming practices on fatty acid composition, inflammatory markers, and metabolomic profiles in adults aged 30-65 years. The study aims to address gaps in understanding the nutritional and health implications of farming practices by comparing postprandial inflammatory and metabolic responses to these diets.

Participants will be randomly assigned to one of two groups and provided with weekly allocations of animal-source foods. Dietary compliance will be assessed through 24-hour dietary recalls and food logs. Blood, urine, and stool samples will be collected at baseline and end of study to measure the primary and secondary outcomes, including:

Red blood cell omega-3 fatty acid levels as a marker of cardiovascular health. A panel of inflammatory markers, including IL-6, TNF-alpha, CRP.

Plasma metabolites such as amino acids, organic acids, and vitamin derivatives.

Lipid profiles (LDL, HDL, VLDL, cholesterol, and triglycerides). Participants will be instructed to consume only the foods provided by the study to ensure dietary control and reduce confounding factors. Biospecimens will be stored for future analysis to examine broader metabolic impacts.

By addressing how different farming practices influence health markers, this study aims to provide evidence-based insights for public health and inform dietary recommendations for sustainable and health-conscious food systems.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 65 years. BMI between 25 and 35 kg/m². Weight stability within the last three months (loss or gain < 4%). Hemoglobin A1C (HbA1C) ≤ 6.4%. Fasting plasma glucose concentration < 126 mg/dL. Ability to understand and communicate in English or Spanish.

Exclusion Criteria:

* Use of medications known to affect study outcomes (e.g., NSAIDs, corticosteroids, anticoagulants) that cannot be discontinued temporarily.

Blood pressure ≥ 140/90 mmHg without physician clearance. Unwillingness to forgo seafood consumption or omega-3 supplement intake during the study.

Alcohol consumption > 14 drinks per week. Tobacco product use within the last three months. Receipt of a COVID vaccine within the last two weeks. Engagement in high-level competitive exercise (e.g., triathlon, marathon, powerlifting).

Diagnosed inflammatory diseases (e.g., autoimmune disorders, coeliac disease, arthritis).

Diagnoses of active malignancy, congestive heart failure, diabetes mellitus, or chronic obstructive pulmonary disease.

Use of antibiotics within the last 60 days. Pregnancy or planning pregnancy within the next month. Lactating women. Allergies to meat or eggs. Inability or unwillingness to comply with the study protocol, including adherence to study visits and dietary requirements.

Dietary preferences that exclude meat or eggs (e.g., vegan, vegetarian, halal). Any condition that, in the opinion of the research team, makes the participant unsuitable for the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only participants who self-identify as male or female are eligible for this study.
Enrollment: 80 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-21 (Actual); Study Completion 2025-09-21 (Actual)

PRIMARY OUTCOMES:
Red Blood Cell (RBC) Omega-3 Fatty Acid Levels | Baseline and 16 weeks (end of intervention).
  Assessment of changes in red blood cell omega-3 fatty acid composition as a marker of cardiovascular health. Blood samples will be collected at baseline and after the 16-week intervention to measure levels using gas chromatography-mass spectrometry (GC and LC/MS).

SECONDARY OUTCOMES:
Metabolomics Profile Analysis | Baseline to Week 16 (End of Study)
  Changes in plasma metabolomic profiles will be assessed to identify variations in metabolites, such as amino acids, organic acids, and vitamin derivatives, associated with the consumption of pastured versus conventional animal products. This analysis will provide insights into the biochemical impacts of dietary interventions on metabolic pathways, inflammation, and overall health. Samples will be analyzed using mass spectrometry for untargeted and/or targeted metabolomics profiling.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Human Nutrition Studies, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Decoded metabolomics data will be shared through public repositories such as Metabolomics Workbench to ensure accessibility. Decoded data on inflammatory biomarkers, gut microbiome profiles, and bloodwork results will be included as supplemental information in peer-reviewed publications resulting from this study.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code

REFERENCES:
- [Background] McAfee AJ, McSorley EM, Cuskelly GJ, Fearon AM, Moss BW, Beattie JA, Wallace JM, Bonham MP, Strain JJ. Red meat from animals offered a grass diet increases plasma and platelet n-3 PUFA in healthy consumers. Br J Nutr. 2011 Jan;105(1):80-9. doi: 10.1017/S0007114510003090. PMID 20807460
- See also: Related Info — https://scholar.google.com/citations?hl=en&user=L5KcySQAAAAJ&view_op=list_works&sortby=pubdate
- See also: Related Info — https://caas.usu.edu/facilities/human-nutrition-studies